CLINICAL TRIAL: NCT05271799
Title: A Randomized, Open-Label, Single-Dose, 2-Period, Crossover Study to Compare Gepotidacin Powder for Oral Suspension With the Adult Tablet Formulation in Healthy Male and Female Participants Aged 18 to 50 Years
Brief Title: A Study to Evaluate Pharmacokinetic, Safety, Tolerability and Relative Bioavailability of Gepotidacin in Healthy Adult Male and Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 207729
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Healthy Volunteers
Keywords: Gepotidacin; Relative Bioavailability; Healthy participants
MeSH Terms: interventions — gepotidacin

STUDY DESIGN:
Intervention Model Description: This is a two periods, crossover study
Masking Description: This is an open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants receiving gepotidacin powder for oral suspension followed by tablet (Experimental)
  Interventions: Drug: Gepotidacin
- Participants receiving gepotidacin tablet followed by powder for oral suspension (Experimental)
  Interventions: Drug: Gepotidacin

INTERVENTIONS:
Drug: Gepotidacin — Gepotidacin will be administered

SUMMARY:
This study is a randomized, open-label, two periods, cross-over pharmacokinetic, safety, tolerability and relative bioavailability of gepotidacin in healthy adult male and female participants of aged 18 to 50 years.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 50 years of age, inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, clinical laboratory tests, vital sign measurements, and 12-lead electrocardiogram results. A participant with a clinical abnormality or laboratory parameters outside the reference range may be included only if the investigator feels and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight more than or equal to (>=) 50.0 kilograms (kg) (110 pound) for males and >=45 kg (99 pound) for females and body mass index within the range 18.5 to 32.0 kilogram per square meters (kg/m^2) (inclusive).
* Male or Female: Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. a. Male participants: Male participants are eligible to participate if they agree to the following during the study intervention period until completion of the follow-up visit: Refrain from donating sperm PLUS, either: Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR Must agree to use contraception/barrier as detailed below: Agree to use a male condom with female partner and should also be advised of the benefit for a female partner to use a highly effective method of contraception, as a condom may break or leak when having sexual intercourse with a woman of childbearing potential (WOCBP) who is not currently pregnant. Agree to use a male condom when engaging in any activity that allows for passage of ejaculate to another person. b. Female participants: A female participant is eligible to participate if she is not pregnant or breastfeeding, and 1 of the following conditions applies: Is not a WOCBP OR Is a WOCBP and using a contraceptive method that is highly effective, with a failure rate of less than (<) 1 percent (%), for at least 30 days prior to dosing until completion of the follow up visit. The investigator should evaluate the potential for contraceptive method failure (e.g., noncompliance, recently initiated) in relationship to the first dose of study intervention. A WOCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) before the first dose of study intervention. The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form and in this protocol.

Exclusion Criteria:

* History or presence of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs, constituting a risk when taking the study intervention, or interfering with the interpretation of data.
* Abnormal blood pressure as determined by the investigator or designee
* Any surgical or medical condition (active or chronic) that may interfere with drug absorption, distribution, metabolism, or excretion of the study intervention, or any other condition that may place the participant at risk, in the opinion of the investigator.
* Positive test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at screening.
* Use of any systemic antibiotic within 30 days of screening.
* Within 2 months before screening, either a confirmed history of Clostridium difficile diarrhea infection or a past positive of Clostridium difficile toxin test.
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert syndrome or asymptomatic gallstones).
* History of drug and/or alcohol abuse within 6 months before screening, as determined by the investigator, or has a positive drug screen at screening or upon admission to the clinic.
* History of sensitivity/hypersensitivity to any of the study drugs, components thereof, or a history of drug or other allergy that, in the opinion of the investigator or the GlaxoSmithKline medical monitor contraindicates their participation.
* History of sensitivity to heparin or heparin-induced thrombocytopenia (if the clinic uses heparin to maintain intravenous cannula patency).
* Impaired sense of taste or smell, in the opinion of the investigator.
* Participants must abstain from taking prescription or non-prescription drugs (except for hormonal contraceptives and/or acetaminophen [up to 2 grams per day]), vitamins, and dietary or herbal supplements, within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to study intervention until completion of the follow-up visit, unless, in the opinion of the investigator and sponsor, the medication will not interfere with the study.
* Participants must abstain from taking QT-prolonging drugs or drugs known to increase the risk of torsades de pointes or the participant is taking a strong cytochrome P450 enzyme 3A4 (CYP3A4) inhibitor within 7 days or 5 half-lives (whichever is longer).
* Previous exposure to gepotidacin within 12 months prior to starting study intervention
* Participant has participated in a clinical trial and has received an investigational product prior to gepotidacin administration within 30 days, 5 half-lives, or twice the duration of the biological effect of investigational product (whichever is longer).
* Participant has participated in a clinical trial with frequent blood sampling and/or sampling blood volumes that in total may reached an extracted blood volume above 7 milliliter per kilogram (mL/kg) (i.e., approximately 500 milliliter (mL) for a 70 kg participant) within the previous 56 days prior to informed consent.
* Presence of hepatitis B surface antigen or positive hepatitis C antibody test result at screening or within 3 months prior to starting study intervention.
* Alanine aminotransferase (ALT) more than (>)1.5 * upper limit of normal (ULN) at screening or check-in.
* Bilirubin >1.5 * ULN (isolated bilirubin >1.5 * ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%) at screening or check-in.
* History of any kidney disease or current or chronic history of impaired renal function as indicated by an estimated creatinine clearance <60 milliliter per minute (mL/min).
* A positive test for human immunodeficiency virus antibody.
* History of regular alcohol consumption within 6 months of screening defined as an average weekly intake of >21 units (or an average daily intake of >3 units) for males or an average weekly intake of >14 units (or an average daily intake >2 units) for females. One unit is equivalent to 270 mL of full-strength beer, 470 mL of light beer, 30 mL of spirits, or 100 mL of wine.
* Urinary cotinine level indicative of smoking or history of regular use of tobacco- or nicotine-containing products within 3 months of screening.
* Clinically significant abnormal findings in serum chemistry, hematology, or urinalysis results obtained at screening or check-in (Day-1).
* Baseline QTcF of >450 milliseconds (msec) at screening or check-in (Day-1).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Periods 1 and 2: Area under the concentration-time curve (AUC) from time zero (pre-dose) extrapolated to infinite time (AUC[0-infinity]) of gepotidacin | Up to 48 hours post dose in each period (each period is 3 days)
  Blood samples will be collected for the concentrations of gepotidacin
Periods 1 and 2: AUC from time zero to the time of the last quantifiable concentration (AUC[0-t]) of gepotidacin | Up to 48 hours post dose in each period (each period is 3 days)
  Blood samples will be collected for the concentrations of gepotidacin
Periods 1 and 2: Maximum observed plasma concentration (Cmax) of gepotidacin | Up to 48 hours post dose in each period (each period is 3 days)
  Blood samples will be collected for the concentrations of gepotidacin

SECONDARY OUTCOMES:
Periods 1 and 2: Number of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 14 days
Periods 1 and 2: Maximum change from Baseline in QT interval corrected with Fridericia's method (QTcF) | Baseline and up to 14 days
Periods 1 and 2: Time to reach maximum observed plasma concentration (Tmax) of gepotidacin | Up to 48 hours post dose in each period (each period is 3 days)
  Blood samples will be collected for the concentrations of gepotidacin.
Periods 1 and 2: Absorption lag time (Tlag) of gepotidacin | Up to 48 hours post dose in each period (each period is 3 days)
  Blood samples will be collected for the concentrations of gepotidacin
Periods 1 and 2: Terminal phase half-life (t1/2) of gepotidacin | Up to 48 hours post dose in each period (each period is 3 days)
  Blood samples will be collected for the concentrations of gepotidacin
Periods 1 and 2: Apparent volume of distribution (Vz/F) of gepotidacin | Up to 48 hours post dose in each period (each period is 3 days)
  Blood samples will be collected for the concentrations of gepotidacin
Periods 1 and 2: Relative bioavailability (Frel) of gepotidacin | Up to 48 hours post dose in each period (each period is 3 days)
  Blood samples will be collected for the concentrations of gepotidacin
Periods 1 and 2: Apparent oral clearance (CL/F) of gepotidacin | Up to 48 hours post dose in each period (each period is 3 days)
  Blood samples will be collected for the concentrations of gepotidacin
Periods 1 and 2: AUC from time zero to 24 hours (AUC[0-24]) of gepotidacin | Up to 24 hours post dose in each period (each period is 3 days)
  Urine samples will be collected for the concentrations of gepotidacin.
Periods 1 and 2: Total unchanged drug (Ae total) of gepotidacin | Up to 48 hours post dose in each period (each period is 3 days)
  Urine samples will be collected for the concentrations of gepotidacin.
Periods 1 and 2: Percentage of the given dose of drug excreted in urine (fe%) of gepotidacin | Up to 48 hours post dose in each period (each period is 3 days)
  Urine samples will be collected for the concentrations of gepotidacin.
Periods 1 and 2: Renal clearance of drug (CLr) of gepotidacin | Up to 48 hours post dose in each period (each period is 3 days)
  Urine samples will be collected for the concentrations of gepotidacin.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com